CLINICAL TRIAL: NCT04311216
Title: Shoulder Instability in Children: Understanding Muscle Activity and Movement Pattern Differences
Brief Title: Shoulder Instability in Children: Muscle Activity and Movement
Status: Completed | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: University of Liverpool (Other); University of Aberdeen (Other); Bournemouth University (Other); Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RL1812
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Injuries; Musculoskeletal Injury; Pediatric ALL; Dislocation, Shoulder; Instability, Joint
MeSH Terms: conditions — Shoulder Injuries; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Shoulder Dislocation; Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shoulder instability participants: Participants with previous a previous episode(s) of shoulder instability
  Interventions: Other: 3D movement analysis with surface electromyography
- Age matched controls (no instability): Participants with no previous a previous episode(s) of shoulder instability
  Interventions: Other: 3D movement analysis with surface electromyography

INTERVENTIONS:
Other: 3D movement analysis with surface electromyography — Single measurement session of 3D movement analysis with surface electromyography for upper limb movements

SUMMARY:
The aim of this study is to identify factors responsible for recurrent shoulder instability in children. Shoulder instability, i.e. complete or partial dislocation of the shoulder joint, is common in children, resulting in pain and disability. Recurrent instability can damage the shoulder joint resulting in the premature development of arthritis.

Rehabilitation approaches are preferred over surgical methods for the growing child e.g. physiotherapy to restore movement and prevent further instability. Existing rehabilitation procedures are based on addressing factors assumed to be responsible for instability e.g. physiotherapists may try to increase shoulder stability by building up the shoulder muscles to compensate for the damaged ligaments. It is evident however that the mechanisms of shoulder instability are not well understood, as failure rates for physiotherapy are high, with 70% - 90% of children continuing to suffer recurrent instability. This is an observational, cross-sectional study of children (aged 8 to 18) presenting with shoulder instability of any origin, traumatic or atraumatic (n=15) and an age-matched sample (n=15) with no history of shoulder problems. Muscle activity and movement pattern differences will be measured using non-invasive 3D motion capture and surface electromyography, to identify factors responsible for instability. Only a single visit to the site will be required (The Orthotic Research & Locomotor Assessment Unit (ORLAU) based at The Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust in Oswestry.).

If investigators better understand the mechanisms associated with instability, physiotherapy interventions to reduce dislocations and disability can be better targeted. If specific patterns of activity associated with instability are identified, these could be addressed through personalised and improved exercise prescription and rehabilitation. Additionally, causes of instability for which physiotherapy may not be appropriate may be identified, therefore ensuring patients are referred to the correct service in a timely manner, improving patient outcomes and allocating physiotherapy resources more appropriately. Participants will be recruited from musculoskeletal/orthopaedic outpatient clinics. This study is funded by the Private Physiotherapy Education Foundation.

ELIGIBILITY:
Inclusion Criteria:

Shoulder instability participants

* Children aged between 8 to 18 years of age
* Subjective reports of instability with additionally symptomatic instability in the clinical assessment criteria below
* Symptomatic instability on clinical assessment in at least one direction, confirmed by a positive clinical finding (apprehension, guarding, laxity) during the sulcus, apprehension or anterior and posterior shift load tests.
* All forms of instability including multidirectional instability, atraumatic and traumatic subluxations and dislocations.
* Children presenting with an initial or recurrent episode of instability
* Children undergoing current management or rehabilitation for their shoulder at the time of the study
* Patients with surgically managed shoulder instability who have since had a further episode of shoulder instability

Age matched controls

- Children aged between 8 to 18 years of age

Exclusion Criteria:

Shoulder instability participants

* Children with co-existing neurological pathologies or deficits
* Surgically managed patients who have not had episodes of instability following the intervention

Age matched controls

* Any previous presentation to a health care professional with a diagnosis of shoulder instability
* Children with a previous shoulder injury within the last 3 months on the arm being assessed that has not resolved
* Children with co-existing neurological pathologies or deficits
* Children who have had a previous surgical intervention on the arm being assessed
* Children currently undergoing or awaiting medical management, diagnostic investigations or rehabilitation on the arm being assessed

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will consist children aged between eight and 18 years of age. The two groups will include children with (shoulder instability participants) and without shoulder instability (age matched contols).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The anonymised final trial dataset and anonymised 3D movement data files will be stored on the Keele University Data repository where they will be assigned a DOI. The anonymised data will be available subject to an appropriate request for research and academic use.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shoulder Instability Participants | Age Matched Controls (no Instability)
Started | 15 | 15
Completed | 13 | 15
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shoulder Instability Participants | Age Matched Controls (no Instability) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (2.9) | 13.3 (3.1) | 13.6 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Shoulder Instability Episodes (Subluxation and Dislocations)
Description: Number of shoulder instability episodes (subluxation and dislocations)
Time Frame: One year
Reporting Status: Not Posted

2. Primary Outcome: Kinematics
Description: Kinematic variables related to the movement tasks - Flexion
Time Frame: On admission
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Shoulder Instability Participants | Age Matched Controls (no Instability)
Number analyzed (Participants) | 15 | 15
degrees
  TH elevation plane | 92 [81 to 102] | 94 [86 to 102]
  TH elevation angle | 133 [122 to 144] | 130 [125 to 134]
  TH rotation | 100 [87 to 113] | 99 [90 to 108]
  TS protraction | 25 [21 to 29] | 24 [21 to 27]
  TS rotation | 39 [37 to 42] | 40 [40 to 44]
  TS tilt | 29 [23 to 36] | 33 [27 to 38]
  GHJ elevation plane | 74 [63 to 85] | 74 [66 to 81]
  GHJ elevation angle | 101 [89 to 112] | 91 [87 to 96]
  GHJ rotation | 89 [79 to 99] | 100 [92 to 108]
  ACJ protraction | 32 [25 to 39] | 34 [29 to 39]
  ACJ rotation | 16 [13 to 20] | 17 [14 to 19]
  ACJ tilt | 31 [28 to 34] | 32 [28 to 36]
  SCJ protraction | 25 [20 to 29] | 24 [21 to 27]
  SCJ elevation | 11 [10 to 12] | 11 [10 to 12]

3. Secondary Outcome: Kinetics
Description: Kinetic variables related to the movement tasks
Time Frame: On admission
Reporting Status: Not Posted

4. Secondary Outcome: Surface Electromyography
Description: Muscle activity patterns related to the movement tasks
Time Frame: On admission
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Shoulder Instability Participants | Age Matched Controls (no Instability)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT04311216/Prot_SAP_000.pdf